CLINICAL TRIAL: NCT07267624
Title: EARLY Antibiotics aDaptation in Ventilator-Acquired-Pneumonia Treatment After Implementation of a Broad-Panel Respiratory Multiplex PCR Test: A Multicenter Randomized Control Trial Conducted In Swiss Intensive Care Units. The EARLY ADAPT Study.
Brief Title: EARLY Antibiotics aDAptation in Severe Pneumonia(The EARLY ADAPT Study)
Acronym: EARLY ADAPT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: BioMérieux (Industry); Hospital Fribourg, Switzerland (Unknown); Hôpital universitaire de Lausanne (Unknown); Hospital of Neuchâtel (Unknown); Centre Hospitalier du Centre du Valais (Other); Hospital Lugano (Unknown)
Responsible Party: Principal Investigator, Christophe Le Terrier, Investigator coordinator and Attending Physician in ICU, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BASEC N° 2024-00369
Record Dates: First submitted 2025-10-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: VAP - Ventilator Associated Pneumonia; Antibiotic; Antibiotic Stewardship; Antibiotic Prescribing for Acute Respiratory-tract Infections; Intensive Care (ICU)
Keywords: ventilator Associated Pneumonia (VAP); antibiotic; PCR multiplex; intensive care; broad spectrum antibiotic; stewardship
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control Group (No Intervention): Care in the control group is based on international guidelines for the management of VAP and carried out in accordance with the local guidelines of each center. This includes respiratory samples with traditional cultures to identify pathogens associated with VAP.
- Intervention Group (Experimental): In the intervention arm, in addition to traditional cultures for identifying pathogens and their resistance, multiplex PCR will be performed on the patient's respiratory samples. Empirical antibiotic therapy will be directly adapted to the results of multiplex PCR according to the guidelines provided.
  Interventions: Device: PCR multiplex BioFire Pneumonia plus

INTERVENTIONS:
Device: PCR multiplex BioFire Pneumonia plus — In the intervention arm, in addition to traditional cultures for identifying pathogens and their resistance, multiplex PCR will be performed on the patient's respiratory samples. Empirical antibiotic therapy will be directly adapted to the results of multiplex PCR according to the guidelines provided.
  Arms: Intervention Group

SUMMARY:
The objective of the study is to determine whether rapid multiplex PCR testing of respiratory samples can reduce exposure to broad-spectrum antibiotics in intensive care unit patients with suspected or confirmed ventilator-associated pneumonia, compared to standard diagnostic methods.

As secondary objectives, the investigators will study antibiotic management and overall antibiotic consumption, as well as escalation or de-escalation events. The investigators will study the potential clinical impact of using multiplex PCR to see if the length of stay in the intensive care unit is reduced, as well as the duration of mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old)
* Hospitalized in intensive care with invasive mechanical ventilation ≥ 48 hours
* Administration of antimicrobial therapy for suspected VAP at the time of inclusion.
* Expected survival > 96 hours.

Exclusion Criteria:

* Enrollment prior to the current trial
* Participation in an interventional study on the management of AMR that has a direct impact on antibiotic therapy practices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the broad-spectrum antibiotic-free hours at day 7 from inclusion | Seven days
  It is defined as the time, measured in hours, that the patient is alive and not treated with broad-spectrum antibiotics (≥ class 4 of ß-lactam according to Weiss et al.) within a period during from the date of randomization to day 7 or earlier if ICU discharge.

SECONDARY OUTCOMES:
Median time (in hours) on broad-spectrum antibiotics during ICU stay. | 28 days
Antibiotic free days defined as the number of days alive without antibiotics at Day 14 and Day 28. | 28 days
Time to antimicrobial switch (time to de-escalation or escalation) measured in hours. | Seven days
Rate of appropriate antimicrobial therapy at the following time points: inclusion, 24h after inclusion and 48h after inclusion. | 48 hours
  I. Appropriate antimicrobial therapy is defined as follows:
  1. Susceptibility of the cultured micro-organisms to the empiric antibiotic regimen.
  2. Narrowest spectrum
  II. Inappropriate antimicrobial therapy is defined as follows:
  1. Not active according to the in-vitro susceptibility testing of the identified pathogen.
  2. Having a spectrum too broad for resistance pattern of the identified pathogen
  3. Known intrinsic resistance of the identified pathogen to the given antibiotic. If no pathogen identified, antibiotic treatment covering Gram-negative rods was considered too broad. These criteria have been selected and adapted by Darie AM et al. Lancet Respir Med. 2022
ICU mortality and hospital mortality at Day 28 | 28 days
Ventilator free-days until Day 28 | 28 days
ICU length of stay | 28 days
Rate of adherence to antimicrobial guidelines at 48h. | 48 hours
  Rate of patients treated following the antimicrobial guidelines provided in the study.

CONTACTS AND LOCATIONS:
Locations (5):
- Switzerland (5):
  - University hospitals of Geneva, Division of Intensive Care, Geneva, Canton of Geneva
  - Dept. of Intensive Care Medicine, University hospital of Lausanne, Lausanne
  - Division of Intensive care, Hospital of Lugano, Lugano
  - Division of Intensive care, Hospital of Neuchâtel, Neuchâtel
  - Division of Intensive care, University hospital of Sion, Sion

IPD SHARING:
Plan to Share IPD: No
Because we would like to publish the IPD before sharing.